CLINICAL TRIAL: NCT02097628
Title: Comparison of Volume- and Pressure- Controlled Ventilation With Laryngeal Mask Airway Guardian in Obese Patients Undergoing Laparoscopic Gynecologic Surgery-A Perspective, Randomized, Blind Trial
Brief Title: Comparison of Two Ventilation Modes With Laryngeal Mask Airway Guardian
Acronym: wang002
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haiyun Wang (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Sponsor-Investigator, Haiyun Wang, M.D., Ph.D., Tianjin Medical University General Hospital
Organization: Tianjin Medical University General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: wang002
Record Dates: First submitted 2014-03-18; First posted 2014-03-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Gynecologic Disease
Keywords: volume controlled ventilation; pressure controlled ventilation
MeSH Terms: conditions — Genital Diseases, Female | interventions — Tidal Volume

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pressure-controlled ventilation (Active Comparator): pressure-controlled ventilation: a peak airway pressure that provided a tidal volume of 8-12ml/kg with an upper limit of 35 centimeter water column, respiratory rate 12-16 times per minute.
  Interventions: Procedure: peak airway pressure
- volume-controlled ventilation (Experimental): volume-controlled ventilation: tidal volume 8-12ml/kg, respiratory rate 12-16 times per minute.
  Interventions: Procedure: tidal volume

INTERVENTIONS:
Procedure: tidal volume — In the volume controlled ventilation group using laryngeal mask airway Guardian,a tidal volume of 8-12ml/kg,respiratory rate12-16bpm.
  Other Names: TV
  Arms: volume-controlled ventilation
Procedure: peak airway pressure — In the pressure controlled ventilation group using laryngeal mask airway Guardian,a peak airway pressure that provides a tidal volume of 8-12ml/kg with an upper limit of 35 centimeter water column,respiratory rate12-16bpm.
  Other Names: airway peal pressure; peak pressure of aieway
  Arms: pressure-controlled ventilation

SUMMARY:
The purpose of this study is to compare volume- and pressure- controlled ventilation with laryngeal mask airway Guardian in obese patients undergoing laparoscopic gynecologic surgery in terms of ventilatory efficacy, airway leak pressure (airway protection), ease-of-use and complications.

DETAILED DESCRIPTION:
The Guardian Laryngeal Mask (Ultimate Medical Pty Ltd, Richmond, Vic, Australia) is a new silicone-based single-use extraglottic airway device that forms a seal with the glottis for ventilation and with the hypopharynx for airway protection, and provides a gastric drainage port. The aim of the following perspective, randomized, blind trial study id to compare how the volume-controlled ventilation and pressure-controlled ventilation modes using the Laryngeal Mask Guardian affect the pulmonary mechanics, the gas exchange and the cardiovascular responses particularly in obese patients undergoing gynecological laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients scheduled to undergo laparoscopic gynecologic surgery under a short general paralysed anesthesia of less than 2 hours (ASA physical status I-II)
* 18 to 65 years of age
* A body mass index <40 kg • m-2

Exclusion Criteria:

* Difficult airway
* Recent history of upper respiratory tract infection and sore throats
* A history of esophageal reflux disease
* Kinesia patients
* Inability to understand the Study Information Sheet and provide a written consent to take part in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
peak pressure | 5 min
  The end-tidal carbon dioxide, the peak pressure, the mean airway pressure, the compliance were continuously monitored during the procedure and they were recorded at T1:just before carbon dioxide insufflation, T2: 30 minutes after carbon dioxide insufflation and T3: 10 minutes after the withdrawal of carbon dioxide. Data on gas exchange (pH、PaCO2、PaO2 ) at T1、T2 and T3 were recorded by artery blood gas analysis.

SECONDARY OUTCOMES:
Blood pressure | intraoperative
  including systolic blood pressure,diastolic blood pressure,mean arterial pressure.
heart rate | intraoperative
  heart rate

OTHER OUTCOMES:
Pharyngolaryngeal complication | 1,24h
  the presence of either sore throat, dysphonia or dysphagia at 1 and 24 h postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Haiyun Wang, M.D.Ph.D., Study Chair — Tianjin Medical University General Hospital